CLINICAL TRIAL: NCT04858230
Title: Pilot Clinical Study to Assess Safety and Feasibility of a New Implantable Device in the Management of Limb Lymphedema
Brief Title: LymphoPilot Test for Limb Lymphedema
Status: Terminated | Phase: Not Applicable | Type: Interventional
Why Stopped: End of shelf life of investigational devices.
Sponsor: Lymphatica Medtech SA (Industry)
Responsible Party: Sponsor
Allocation: Not Applicable | Model: Single Group | Masking: None | Purpose: Device Feasibility
Other Study IDs: LymphoPilot
Record Dates: First submitted 2021-04-13; First posted 2021-04-26 (Actual); Last update posted 2025-03-07 (Actual); Status verified 2025-03

CONDITIONS: Lymphedema, Secondary; Lymphedema of Upper Limb; Lymphedema Arm; Lymphedema of Leg; Lymphedema, Lower Limb
Keywords: lymphedema
MeSH Terms: conditions — Lymphedema; Neoplasm Metastasis

STUDY DESIGN:
Oversight: Data Monitoring Committee: Yes | FDA-regulated Drug: No | FDA-regulated Device: No | US Export: No

ARMS (1):
- LymphoPilot (Experimental): Patient will be implanted with the medical device under investigation, LymphoPilot, through a surgical procedure performed in loco-regional or general anesthesia. Lymphedema outcomes will be monitored for 8 weeks after implantation and compared to baseline values before device implantation. Safety data will be collected throughout the study.
  Interventions: Device: LymphoPilot

INTERVENTIONS:
Device: LymphoPilot — LymphoPilot is an investigational medical device composed of an implanted part (pump, drainage catheter and output catheter), implanted in the subcutaneous tissue of the arm or of the leg and draining excess fluids to the supraclavicular or abdominal subcutaneous tissue, where fluids are naturally reabsorbed by the healthy lymphatic and venous system. The implanted part is activated and controlled via a wearable device.
  The subcutaneous implantation of the device is performed in loco-regional or general anesthesia, in ambulatorial settings, and the patient is dismissed from the hospital on the same day of the procedure.
  Patients will wear the external controller continuously throughout the study, except 30 minutes per day, to allow taking a shower/bath. The implanted device will be removed with a surgical procedure in local anesthesia 8 weeks after device implantation.

SUMMARY:
The present study is a first-in-man, single arm, open-label, single center study to assess feasibility and safety of a novel implantable device, LymphoPilot, in patients suffering from secondary upper limb or lower lymphedema.

DETAILED DESCRIPTION:
The study consists in a first-in-man clinical investigation for LymphoPilot, an investigational implantable medical device. LymphoPilot is composed of an implanted part and an external wearable device. The implanted part (pump, drainage catheter and output catheter), is implanted in the subcutaneous tissue of the arm or leg and drains excess fluids to the supraclavicular or abdominal subcutaneous tissue, where fluids are naturally reabsorbed by the healthy lymphatic and venous system. The external part consists in a wearable controller used to activate the implanted pump.

The subcutaneous implantation of the device is performed in loco-regional or general anesthesia, in ambulatorial settings, and the patient is dismissed from the hospital on the same day of the procedure.

The device is activated in the postoperative room by placing the external wearable device on patient's limb, in proximity of the implanted pump. Patients are required to wear the external controller continuously throughout the study, except 30 minutes per day, to allow taking a shower/bath.

Follow-up visits are planned 1, 4 and 8 weeks after device implantation. The implanted device is removed with a surgical procedure in local anesthesia 8 weeks after device implantation, and 2 additional follow-up visits are planned after device removal.

ELIGIBILITY:
Inclusion Criteria:

* Female patients, 18 years and older
* Patients with unilateral secondary upper or lower limb lymphedema.

Exclusion Criteria:

* Active cellulitis/infection
* Lymphedema associated with active cancer requiring chemotherapy or radiotherapy
* Motor and sensitive neurological deficiency
* Post-operative edema (i.e. acute edema following breast cancer related surgery)
* Any contraindication to surgery or to loco-regional or general anesthesia
* Patient participating in any other clinical study
* Patient unable to provide informed consent
* Patient with pacemaker
* Pathologies associated with an overload of the cardiac system
* Poor wound healing
* Pregnancy or breastfeeding
* Known intolerance to implantable devices
* Known allergies to silicone
* Patient needing magnetic therapy
* Any other condition that according to the principal investigator makes the patient unsuitable for the participation in the trial
* Patient refusing to receive information about incidental findings on her health status discovered during the clinical investigation
* L-Dex score lower than 6.5 at screening

Min Age: 18 Years | Sex: Female | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Enrollment: 12 (Actual)
Dates: Start 2021-09-08 (Actual); Primary Completion 2023-09-30 (Actual); Study Completion 2023-09-30 (Actual)

PRIMARY OUTCOMES:
Occurrence, frequency and severity of device-related adverse events | From enrollment until final visit, 4 weeks after device removal.
  Occurrence, frequency and severity of device-related adverse events are used to evaluate device safety

SECONDARY OUTCOMES:
Device functionality evaluated via ultrasound imaging | At day 1 (implant surgery), day 7, day 28 and day 56
  Ultrasound imaging is used to verify fluid flow in the implanted catheters
Limb volume | At day 0 (baseline), day 7, day 28, day 56, day 66, day 84
  Arm or leg volume evaluated by tape measure and by perometer
L-Dex score | At day 0 (baseline), day 7, day 28, day 56, day 66, day 84
  L-Dex score is measured via bioimpedance spectroscopy
Upper extremity function | At day 0 (baseline) and at day 56
  The Quick Disability of Arm, Shoulder, Hand Questionnaire (DASH) is used to evaluate upper extremity function
Lower extremity function | At day 0 (baseline) and at day 56
  The Lower Extremity Functional Scale (LEFS) is used to evaluate lower extremity function
Physical functioning evaluated via validated SF-36 questionnaire | At day 0 (baseline) and at day 56
  The Short Form-36 (SF-36) questionnaire is used to evaluate patient's physical functioning.
  Scoring scale: 0 to 100%, where the highest percentage represents the best outcome.
Role limitations due to physical health evaluated via validated SF-36 questionnaire | At day 0 (baseline) and at day 56
  The Short Form-36 (SF-36) questionnaire is used to evaluate patient's role limitations due to physical health.
  Scoring scale: 0 to 100%, where the highest percentage represents the best outcome.
Role limitations due to emotional problems evaluated via validated SF-36 questionnaire | At day 0 (baseline) and at day 56
  The Short Form-36 (SF-36) questionnaire is used to evaluate patient's role limitations due to emotional problems.
  Scoring scale: 0 to 100%, where the highest percentage represents the best outcome.
Energy/fatigue evaluated via validated SF-36 questionnaire | At day 0 (baseline) and at day 56
  The Short Form-36 (SF-36) questionnaire is used to evaluate patient's energy/fatigue.
  Scoring scale: 0 to 100%, where the highest percentage represents the best outcome.
Emotional well-being evaluated via validated SF-36 questionnaire | At day 0 (baseline) and at day 56
  The Short Form-36 (SF-36) questionnaire is used to evaluate patient's emotional well-being.
  Scoring scale: 0 to 100%, where the highest percentage represents the best outcome.
Social functioning evaluated via validated SF-36 questionnaire | At day 0 (baseline) and at day 56
  The Short Form-36 (SF-36) questionnaire is used to evaluate patient's social functioning.
  Scoring scale: 0 to 100%, where the highest percentage represents the best outcome.
Pain evaluated via validated SF-36 questionnaire | At day 0 (baseline) and at day 56
  The Short Form-36 (SF-36) questionnaire is used to evaluate patient's pain. Scoring scale: 0 to 100%, where the highest percentage represents the best outcome.
General health evaluated via validated SF-36 questionnaire | At day 0 (baseline) and at day 56
  The Short Form-36 (SF-36) questionnaire is used to evaluate patient's general health.
  Scoring scale: 0 to 100%, where the highest percentage represents the best outcome.
Quality of life evaluated via validated LYMQOL-leg questionnaire | At day 7 and at day 56
  The Lymphedema Quality of Life Questionnaire for leg Lymphedema (LYMQOL-LEG) questionnaire is used to evaluate assessing problems in functioning in patients with lower limb lymphedema.
  Scoring scale: 0-10, where highest scores represent the best outcome.
Quality of life evaluated via validated LYMPH-ICF-UL questionnaire | At day 7 and at day 56
  The Lymphedema Functioning, Disability and Health Questionnaire for Upper Limb Lymphedema (LYMPH-ICF-UL) questionnaire is used to evaluate assessing problems in functioning in patients with upper limb lymphedema.
  Scoring scale: 0-100, where highest scores mean a worse outcome.
Ease of use of the device | At day 7 and at day 56
  Device usability evaluated via dedicated survey

CONTACTS AND LOCATIONS:
Overall Officials: Lucia Mazzolai, Prof., Principal Investigator — CHUV
Locations (1):
- Angiology Service - Centre Hospitalier Universitaire Vaudois (CHUV), Lausanne, Canton of Vaud, Switzerland

IPD SHARING:
Plan to Share IPD: No

REFERENCES:
- [Background] Mazzolai L, Triacca V, Brochu-Vez MJ, Boucard V, Aberle M, Chaplet V, Ferrari V, Deglise S, Pisano M, Staubli S. Advancing women's health with a pioneering implant to treat breast cancer related lymphedema. Eur J Intern Med. 2025 May;135:64-73. doi: 10.1016/j.ejim.2025.01.027. Epub 2025 Feb 12. PMID 39939264